CLINICAL TRIAL: NCT02571959
Title: Pharmacokinetic Study of the Amoxicillin / Clavulanic Acid Association to Optimize Dosage Among Obese Adults (PHACO)
Brief Title: Pharmacokinetic Study of the Association of Amoxicillin / Clavulanic Acid to Obese Adults
Acronym: PHACO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMEA 046
Record Dates: First submitted 2015-04-14; First posted 2015-10-08 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Obesity
Keywords: Obesity; Pharmacology; Amoxicillin-Potassium Clavulanate Combination
MeSH Terms: conditions — Obesity | interventions — Amoxicillin-Potassium Clavulanate Combination; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- amoxicillin and clavulanic acid (Experimental): All volunteers receive a dose of amoxicillin and clavulanic acid
  Interventions: Drug: amoxicillin and clavulanic acid

INTERVENTIONS:
Drug: amoxicillin and clavulanic acid — Day 1 : a dose of amoxicillin and clavulanic acid 1g / 200mg will be intravenously administered
  Other Names: AMOXICILLINE / acide clavulonique SANDOZ
Drug: amoxicillin and clavulanic acid — Day 2 : a dose of amoxicillin and clavulanic acid 1g / 125mg will be administered by oral route
  Other Names: AMOXICILLINE / acide clavulonique SANDOZ

SUMMARY:
Description of the pharmacokinetic parameters of the amoxicillin / clavulanic acid to healthy voluntary obese after oral and intra venous administration Determination of the pharmacokinetic parameters of amoxicillin / clavulanic acid obtained from plasmatic concentrations of intravenous injection (IV) and oral administrations. The criterion of evaluation allowing to answer our main objective corresponds to the parameters estimated by the pharmacokinetic model of the concentrations obtained from the data IV and by the pharmacokinetic model of the concentrations obtained from the oral data. The following pharmacokinetic parameters will be considered at every obese volunteer's for both molecules (amoxicillin and clavulanic acid) from the concentrations by pharmacokinetic analysis of population.

The main evaluation criteria are PK parameters of amoxicillin / clavulanic:

* Cl, systematic plasmatic clearance
* Vd, volume of distribution
* ASC 0-oo, area under the curve time - concentration
* T1/2, half-life time
* F, bioavailability after oral administration
* Ka, constant of speed of absorption

DETAILED DESCRIPTION:
Main objective Description of the pharmacokinetic parameters of the amoxicillin / clavulanic acid to healthy voluntary obese after oral and intra venous administration

Secondary objectives

* Define dosage plans optimized with the antibiotic treatment to the obese subject
* Ensure an adequacy of the treatment with the related infection
* Formulate recommendations of dosage adaptations for a better individualization of treatments, by estimating several plans of doses by simulation to reach various PK/PD goals according to different theoretical MIC

Methodology

The pharmacokinetic analysis will be realized by approach of population allowing the estimation of the average parameters of amoxicillin and clavulanic acid as well as the interpersonal variability after an administration IV and an oral administration. Parameters's population and their variability will be estimated with the SAEM algorithm implemented in the software Monolix ( www.lixoft.eu ).

For the main objective, PK parameters PK of amoxicillin and clavulanic acid will be determined to day 1 and day 2. They will be described by means of indicators of position (average and median) and of dispersal (standard deviations, quartiles).

For secondary objectives, the profiles concentration/time of 1000 obese subjects will be determined by Monte Carlo method from PK parameters estimated at the balance by the model. For every feigned profile, the time during which the plasmatic concentration of amoxicillin and clavulanic acid is superior to a panel of theoretical MIC will be calculated by means of curves concentration - time determined for each of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary obese
* Body mass index upper to 30 kg/m2
* Age from 18 to 65 years
* Signed free and lit consent
* Possible participation according to the national file of the volunteers of the French Ministry of Health.
* Volunteers affiliated to the Social Security

Exclusion Criteria:

* Pregnancy
* Evolutionary pregnancy or feeding
* Allergy in ß-lactamines (nettle rash, oedema of Quincke)
* Digestive intolerance with amoxicillin / clavulanic acid
* Infection by the virus of the HIV ( positive Ac anti HIV)
* Infection by the virus of the hepatitis B ( positive Ag Hbs)
* Infection by the virus of the hepatitis C ( positive Ac anti VHC)
* Hepatic cirrhosis at the Child-Pugh C stage(stadium)
* Biological parameters:
* Polynucléaires neutrophiles 750 / mm3
* Haemoglobin 8g / dL
* Patellets 60 000 / mm3
* Creatinin clearance, according to MDRD, DFG 50 mL / min / 1,73m2
* ASAT or ALAT > 3 times the superior limit of the normal (LSN)
* Phosphatase alkaline > 3 LSN
* Total Bilirubine > 3 LSN
* Lipase > 3 LSN
* Factor V < 50 %
* Alcoholism chronicles (consumption superior to 30 g of alcohol a day, amount to 3 glasses of wine)
* Significant anomaly of the electrocardiogram, in particular QTc > 450 msec
* Subject susceptible not to respect the modalities of the study
* Drug addiction intra venous
* Any medical conditions which according to the judgment(sentence) of the investigator would may interfere with the moderate pharmacokinetic parameters
* People placed under legal protection
* Histories of bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2015-10-13 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Systematic plasmatic clearance (Cl) | 1 day

SECONDARY OUTCOMES:
Area under the curve time - concentration (AUC 0-oo) | 1 day
Half-life time (T1/2) | 1 day
Volume of distribution (Vd) | 1 day
Bioavailability after oral administration (F) | 1 day
Constant of speed of absorption (Ka) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Ambroise Pare, Boulogne, France